CLINICAL TRIAL: NCT05420350
Title: A Randomized, Prospective, Double-Blind, Placebo-Controlled, Pilot Study to Assess the Effectiveness of a Combination of Lamotrigine and Bupropion to Treat Meniere's Disease
Brief Title: Lamotrigine and Bupropion for Meniere's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dent Neuroscience Research Center (Other)
Collaborators: Cures Within Reach (Other); Dent Family Foundation (Unknown)
Responsible Party: Principal Investigator, Lixin Zhang, Medical Director of the Dizziness and Balance Center, Dent Neuroscience Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DBTC-003
Record Dates: First submitted 2022-05-26; First posted 2022-06-15 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Meniere Disease; Ménière's Vertigo; Vertigo, Intermittent; Vertigo, Aural
Keywords: Lamictal; Lamotrigine; Anticonvulsant; Meniere's Disease; Vertigo attack; Dizziness; Vestibular disorder; Wellbutrin; Bupropion
MeSH Terms: conditions — Meniere Disease; Vertigo; Dizziness; Vestibular Diseases | interventions — Lamotrigine; Bupropion; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Subjects randomized to receive lamotrigine and bupropion or matching placebo randomized 1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lamotrigine and Bupropion (Active Comparator): Lamotrigine will be taken orally for a duration of 28 weeks, consisting of a six-week titration, 20-week study period, and two-week taper. Possible doses are 25mg one a day, 50mg once a day, 50mg twice a day, 75mg twice a day during titration; 125mg twice a day for the study period; and 125mg once a day during the two-week taper. Patients who discontinue at any point of the study will have a two-week taper of lamotrigine.
  Bupropion will be taken orally for the duration of 20 week at the dosage of 100mg twice a day.
  Interventions: Drug: Lamotrigine and Bupropion
- Placebo (Placebo Comparator): The placebo will match the lamotrigine and bupropion dosage, frequency, and duration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lamotrigine and Bupropion — Lamotrigine-oral pill taken once or twice a day with varying dosage per study timeline Bupropion-oral pill 100mg taken twice a day
  Other Names: Lamictal; Lamictal ODT; Lamictal XR; Wellbutrin XL; Wellbutrin SR; Forfivo XL
  Arms: Lamotrigine and Bupropion
Drug: Placebo — Oral pill matched with lamotrigine to be taken once or twice a day per study timeline Oral pill matched with bupropion to be taken twice a day
  Other Names: Microcrystalline cellulose
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled clinical trial to assess whether treatment with lamotrigine and bupropion is more effective than placebo to reduce definitive Meniere's vertigo attacks (DMVA) and dizziness in patients with Meniere's disease. Thirty four participants will be randomized to treatment or placebo groups. Each participant will take part in the trial for 34 weeks, or approximately 9 months.

DETAILED DESCRIPTION:
Participants begin with a 4 week lead-in after screening to determine the frequency and severity of vertigo they are experiencing. Participants continue to track their vertigo episodes throughout the study. At Visit 2, if eligible, participants begin the titration of lamotrigine or matching placebo. Participants are on the full dose of lamotrigine/placebo for 8 weeks, and then begin taking bupropion or matching placebo along with lamotrigine or matching placebo for 12 weeks. At Week 27, participants are tapered off lamotrigine/placebo and stop taking bupropion/placebo. Participants have an in-person visit approximately once a month over 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, male and female aged 18 years or older
* Diagnosis of definitive unilateral Meniere's disease according to the AAO-HNS 1995 criteria, confirmed by an ENT or qualified medical professional
* Be experiencing active vertigo
* Be in good general health as evidenced by medical history or, otherwise, have all other co-existing medical or psychiatric conditions stable, and or no greater than moderate in severity, as determined by the PI
* Females of childbearing potential must use at least two forms of acceptable contraception, or remain abstinent; male participants must be willing to use condoms or other methods to ensure effective contraception with a partner
* Be willing to comply with all study procedures and availability for the duration of the study
* Be able to provide informed written consent, including agreement to privacy language either within the informed consent or in ancillary documents compliant with Health Insurance Portability and Accountability Act (HIPAA) before the initiation of any study-related procedures

Exclusion Criteria:

* A diagnosis of bilateral Meniere's disease according to the AAO-HNS 1995 criteria, confirmed by an ENT or qualified medical professional
* Be pregnant or lactating
* Have active migraine-associated vertigo
* Not be able to accurately identify and report episodes of vertigo
* Diagnosis of any other neuro-otologic disease or major vestibular abnormality found during screening that could confound the evaluation of Meniere's symptoms
* Have a history of intolerance or sensitivity to lamotrigine
* Previously failed the study drug
* Received an intratympanic gentamicin injection(s) or endolymphatic sac surgery within in the last year
* Have a family history of unexplained deafness
* Have any current diseases or conditions that may be associated with an altered perception of processing stimuli
* Have a history of substance abuse within the preceding 6 months prior to screening
* Have non-vertiginous dizziness (orthostatic or panic disorder) unless it could be clearly differentiated from Meniere's attacks by the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in Ménière's vertigo attack frequency between groups | Duration of lead-in to completion at week 30
  Number of Definitive Ménière's Vertigo attacks (DMVA), Number of Dizziness Days and overall dizziness severity during each 4-week of titration, and treatment compared to the 4-week lead-in phase. Vertigo ratings will be collected on a daily symptom diary throughout the study. DMVA is defined as vertigo for more than 20 minutes and corresponds to a vertigo rating of 3 or 4 on the daily symptom diary. A Dizziness Day is defined as vertigo rating of 1, 2, 3 or 4 on the daily symptom diary. Dizziness severity is the sum of all ratings (0-4) during each 4-week period.
Change in Ménière's vertigo attack frequency lamotrigine alone compared to lamotrigine and bupropion | Week 1 to Week 27
  Number of Definitive Ménière's Vertigo attacks (DMVA), Number of Dizziness Days and overall dizziness severity during each 4-week of treatment of lamotrigine alone and treatment of bupropion and lamotrigine.Vertigo ratings will be collected on a daily symptom diary throughout the study. DMVA is defined as vertigo for more than 20 minutes and corresponds to a vertigo rating of 3 or 4 on the daily symptom diary. A Dizziness Day is defined as vertigo rating of 1, 2, 3 or 4 on the daily symptom diary. Dizziness severity is the sum of all ratings (0-4) during each 4-week period.

SECONDARY OUTCOMES:
Changes in patients' self-assessment of dizziness | Baseline (Week 1) and Visit 8 (Week 27)
  Between groups comparisons of Dizziness Handicap Inventory (DHI) at Week 27 compared to the baseline visit at the end of the lead-in phase. DHI at baseline compared to evaluation at end of treatment.
  Scores range from 0-100 with higher scores meaning more severe dizziness handicap
Changes in patients' self-assessment of overall affect of symptoms | Baseline (Week 1) and Visit 8 (Week 27)
  Between groups comparisons of Ménière's Disease Patient-Oriented Symptom-Severity Index (MDPOSI) at Week 27 compared to the baseline visit at the end of the lead-in phase. MDPOSI at baseline compared to evaluation at end of treatment.
  Scores range from 0-80 with higher numbers indicating more frequent and severe symptoms.
Changes in patients' self-assessment of symptom impact on daily life function | Baseline (Week 1) and Visit 8 (Week 27)
  Between groups comparisons of Ménière's Disease Self-Assessment (MDSA) at Week 27 compared to the baseline visit at the end of the lead-in phase. MDSA at baseline compared to evaluation at end of treatment.
  Scores range from 1-6 with higher numbers representing Ménière's Disease symptoms having a greater affect on the patient's ability to function in daily life.
Changes in patients' self-assessment of depression | Baseline (Week 1) and Visit 8 (Week 27)
  Between groups comparisons of Patient Health Questionnaire-9 (PHQ-9) at Week 27 compared to the baseline visit at the end of the lead-in phase. PHQ-9 at baseline compared to evaluation at end of treatment.
  Scores range from 0-27 with higher numbers meaning more severe depression.
Changes in patients' self-assessment of anxiety | Baseline (Week 1) and Visit 8 (Week 27)
  Between groups comparisons of General Anxiety Disorder-7 (GAD-7) at Week 27 compared to the baseline visit at the end of the lead-in phase. GAD-7 at baseline compared to evaluation at end of treatment.
  Scores range from 0-21 with higher numbers meaning more severe anxiety.

OTHER OUTCOMES:
Change in patients' tinnitus from baseline to the end of treatment. | Baseline (Week 1) and Visit 8 (Week 27)
  Between groups comparisons of Tinnitus Handicap Index (THI) at Week 27 compared to the baseline visit at the end of the lead-in phase. THI at baseline compared to evaluation at end of treatment.
  Score range from 0-100 with higher numbers representing a more severe tinnitus handicap.
Change in patients' hearing loss from baseline to the end of treatment. | Baseline (Week 1) and Visit 8 (Week 27)
  Between groups comparisons of hearing loss at Week 24 compared to the baseline visit at the end of the lead-in phase. Hearing loss measured based off the pure-tone average at 500 Hz, 1000 Hz, 2000 Hz, and 3000 Hz measured in dB from audiometric report taken at Visit 1 and Visit 8.

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Zhang, MD, PhD, Principal Investigator — Dent Neurologic Institute
Locations (1):
- Dent Neurologic Institute, Amherst, New York, United States